CLINICAL TRIAL: NCT01197807
Title: Newborn Resuscitation: A Randomized Controlled Trial of Oronasopharyngeal Suction Versus Simple Nose and Mouth Wiping in Term Newborns
Brief Title: Oronasopharyngeal Suction Versus Simple Nose and Mouth Wiping in Term Newborns
Acronym: TermWIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John Kelleher, MD, Fellow Instructor, Department of Pediatrics, Division of Neonatology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB Neo 001
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy, Childbirth and the Puerperium; Resuscitation
Keywords: Suctioning; Wiping; Neonate; Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bulb suctioning (Active Comparator): Bulb suctioning of mouth and nose immediately after delivery
  Interventions: Procedure: Bulb Suctioning
- Wiping (Active Comparator): Gentle wiping of mouth then nose with soft cloth
  Interventions: Procedure: Wiping

INTERVENTIONS:
Procedure: Bulb Suctioning — Bulb suctioning of the mouth then the nose immediately following delivery
  Arms: Bulb suctioning
Procedure: Wiping — Gentle wiping of mouth then nose with a soft cloth immediately following delivery
  Arms: Wiping

SUMMARY:
Until recently, bulb or catheter oronasopharyngeal suctioning (ONPS) of all the infants, including vigorous infants in the delivery room, has been featured as a standard of newborn care. The 5th edition of the Newborn Resuscitation Program (NRP) has minimized the recommendation for routine suctioning of infants following delivery, provided they are not depressed or in need of immediate resuscitation. However, this new alternative recommendation was based on a small randomized trial and other lower level evidence rather than evidence from larger trials. The NRP Textbook cautions against vigorous suctioning because of the resultant apnea or bradycardia. Furthermore, suctioning may delay other more important steps of resuscitation. Thus, it is necessary to compare the alternative recommended practice, i.e. simple wiping of the mouth, to determine if it has equivalent efficacy and a favorable side effect profile compared to suctioning.

ELIGIBILITY:
Inclusion Criteria:

* Inborn neonates at the UAB hospital with gestational age greater than or equal to 35 weeks.

Exclusion Criteria:

* Major birth anomalies or where a decision to institute comfort care only has been made antenatally
* Significant resuscitation efforts are anticipated prior to delivery
* Nonvigorous infants with meconium stained amniotic fluid

Ages: 1 Minute to 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 506 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Mean respiratory rate over the first 24 hours of life | 24 hours after birth
  Respiratory rates measured every 8 hours during the first 24 hours after birth

SECONDARY OUTCOMES:
Apgar Scores at one minute of age | 1 minute of age
  Independent assignment of Apgar Scores at one minute of age
Number of newborns with tachypnea | 24 hours
  Number of newborns with tachypnea as defined by respiratory rate greater than 60 breaths per minute
Need for delivery room resuscitation | 1 hour after birth
  Need for delivery room resuscitation including suctioning, intubation, positive pressure ventilation, chest compressions, and/or medication
Admission to the Neonatal Intensive Care Unit | 1 hour after birth
  Needing admission to the Neonatal Intensive Care Unit
Oxygen saturations prior to discharge from hospital | 5 days of age
  Measurements of oxygen saturations in the well baby nursery prior to discharge home
Apgar score at 5 minutes of age | 5 minutes of age
  Independent assignment of Apgar score at 5 minutes of age

CONTACTS AND LOCATIONS:
Overall Officials: John Kelleher, MD, Principal Investigator — University of Alabama at Birmingham; Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Kelleher J, Bhat R, Salas AA, Addis D, Mills EC, Mallick H, Tripathi A, Pruitt EP, Roane C, McNair T, Owen J, Ambalavanan N, Carlo WA. Oronasopharyngeal suction versus wiping of the mouth and nose at birth: a randomised equivalency trial. Lancet. 2013 Jul 27;382(9889):326-30. doi: 10.1016/S0140-6736(13)60775-8. Epub 2013 Jun 3. PMID 23739521